CLINICAL TRIAL: NCT00826449
Title: Phase I-II Study of Dasatinib and Erlotinib in Non-Small Cell Lung Cancer
Brief Title: Dasatinib and Erlotinib in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0353; NCI-2012-01653 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Advanced Solid Tumors; Advanced Cancer; Non-Small Cell Lung Cancer; NSCLC; Solid Tumor Malignancy; Dasatinib; BMS-354825; Sprycel®; Erlotinib; Erlotinib hydrochloride; Tarceva; OSI-774
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Dasatinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase I (Experimental): Dasatinib + Erlotinib
  Interventions: Drug: Dasatinib; Drug: Erlotinib

INTERVENTIONS:
Drug: Dasatinib — Starting dose of 70 mg by mouth daily for 21 day cycle.
  Other Names: BMS-354825; Sprycel®
Drug: Erlotinib — 150 mg by mouth daily every 21 day cycle.
  Other Names: Erlotinib hydrochloride; Tarceva; OSI-774

SUMMARY:
The goal of the Phase I portion of this study is to find the highest tolerable dose of the combination of dasatinib and erlotinib hydrochloride that can be given to patients with advanced solid tumors.

The goal of the Phase II portion of this study is to learn if this combination is effective when given to patients with non-small cell lung cancer.

The safety of this combination will be studied in both phases.

DETAILED DESCRIPTION:
The Study Drugs:

Dasatinib is designed to decrease the activity of one or more proteins that are responsible for the uncontrolled growth of tumor cells. This may cause the tumor cells to die.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells. Blocking the protein may control tumor growth and survival. This may stop tumors from growing.

Study Groups:

If you are found to be eligible to participate in this study, you will be assigned to a study group based on when you joined this study. Up to 6 groups of 3-6 participants each will be enrolled in the Phase I portion of the study, and up to 35 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of dasatinib you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of dasatinib. Each new group will receive a higher dose of dasatinib than the group before it, if no intolerable side effects were seen. If intolerable side effects are seen, the next group of participants may receive the same dose level or a lower dose level. This will continue until the highest tolerable dose of dasatinib is found.

If you are enrolled in the Phase II portion, you will receive highest tolerated dose level of dasatinib that was found in the Phase I portion.

All participants will receive the same dose level of erlotinib hydrochloride. If the doctor thinks it is needed, the dose level may be lowered.

Study Drug Administration:

If you are in Phase I, on Day -3 of Cycle 1 (3 days before your first dose of study drugs), you will take erlotinib hydrochloride by mouth. On Days 1-19 of Cycle 1, you will be take dasatinib and erlotinib hydrochloride by mouth once a day. On Days 20 and 21 of Cycle 1, you will only take dasatinib by mouth once a day. Every day of Cycles 2 and beyond, you will take dasatinib and erlotinib hydrochloride by mouth once a day.

If you are in Phase II, every day you will take dasatinib and erlotinib hydrochloride by mouth once a day.

Each cycle is 21 days.

Erlotinib hydrochloride and dasatinib should be taken together at the same time every day. The tablets must be swallowed whole and may not be broken. The tablets should be taken with 1 cup (about 8 ounces) of water. Dasatinib and erlotinib hydrochloride should be taken 1 hour before or 2 hours after meals or any other drugs, and should not be taken with grapefruit juice. The entire dose must be taken at 1 time. If you vomit within 30 minutes of swallowing the tablets, the dose may be replaced if the tablets can be seen and counted. If you are currently taking St. John's Wort, you should stopping taking if for at least 5 days before taking dasatinib.

Study Visits:

At Week 1 of Cycle 1, your vital signs and weight will be measured.

At the end of Week 3 of every cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a performance status evaluation.
* Blood (about 1 tablespoon) will be drawn for routine tests
* The amount of oxygen in your blood will be measured by a pulse oximeter.
* You will have a chest x-ray to check the status of the disease.
* You will be asked if you have experienced any side effects and to list any drugs you may be taking.
* Women who are able to become pregnant must have a negative blood (about 1-2 teaspoons) or urine pregnancy test.

At the end of Week 3 of Cycles 1 and 3, you will also have an ECG.

At the end of Week 3 of every other cycle (Cycles 2, 4, 6, and so on), you will also have a chest CT scan or a whole body PET/CT (if necessary) to check the status of the disease.

Phase I PK Testing:

If you are in Phase I, you will have blood (about 2 teaspoons each time) drawn for PK testing.

* On Day -3 of Cycle 1, blood will be drawn 5 different times.
* On Days -2, -1, and 1 of Cycle 1, blood will be drawn 1 time.
* On Day 19 of Cycle 1, blood will be drawn 5 times.
* On Days 20, 21, and 22 of Cycle 1, blood will be drawn 1 time.

Length of Study:

You may stay on study for as long as you are benefitting. You will be taken off study if you experience intolerable side effects or the disease gets worse.

End-of-Study Visit:

At the end of your study participation, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a performance status evaluation.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* The amount of oxygen in your blood will be measured.
* You will have a chest x-ray to check the status of the disease.
* You will have an ECG.

If you are taken off study due to unacceptable side effects, you will be called and asked about any side effects until the side effect gets better or becomes stable.

Long-Term Follow-Up:

After the end-of-study visit, you will be contacted every 3-4 months for 1 year to collect information about how you are doing. You (or your family members or designees) may be contacted by telephone or during clinic visits. If you are called, this will take about 5 minutes.

This is an investigational study. Dasatinib is FDA approved and commercially available for the treatment of acute lymphoid and chronic myeloid leukemia. Erlotinib hydrochloride is FDA approved and commercially available for the treatment of non-small cell lung cancer. The use of this combination in this study is investigational.

Up to 59 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced malignancy that is appropriate for systemic therapy without curative intent.
2. Patients must provide verbal and written informed consent indicating they are aware of the investigational nature of the study. Parental consent and patient assent is required for those aged 16-17.
3. Patients must be at least 16 years of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. Adequate hematologic, hepatic, and renal function as follows: creatinine < 1.5 x the institutional upper limit of normal (ULN), total bilirubin < 2.0 x ULN, AST and ALT < 2.5 x ULN, absolute granulocytes >/= 1500/mm^3; platelets >/= 75,000 mm^3; hemoglobin >/= 10 g/dL.
6. Serum potassium, magnesium, and phosphate within the institutional limits of normal. Patients with low potassium, phosphate, or magnesium levels may be repleted to allow for protocol entry.
7. Serum calcium >/= the institutional limits of normal. Patients with low calcium levels may be repleted to allow for protocol entry.
8. Ability to take oral medication (dasatinib and erlotinib must be swallowed whole)
9. Patients-both males & females-w/reproductive potential must agree to use an adequate method of contraception to include hormonal contraceptives (birth control pills, injections, implants), intrauterine device (IUD), barrier contraceptive with spermicide, and/or abstinence throughout the study & for at least 4 wks after the study drugs are stopped. Females w/ reproductive or childbearing potential include any female who has experienced menarche & who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal
10. -Continued from Inclusion #9 - [defined as amenorrhea >/=12 consecutive mths;or women on hormone replacement therapy (HRT) w/ documented serum follicle stimulating hormone (FSH) level > 35 milli-International unit (mIU)/mL]. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
11. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 72 hours prior to the start of study drug administration.
12. Asymptomatic brain metastases with prior cranial irradiation or resection are acceptable if there is no bleeding, no midline shift, and no need for steroids or anti-convulsants. Asymptomatic brain metastasis without prior treatment are acceptable if the largest lesion is less than 7 mm in diameter, there is no bleeding, midline shift, nor need for steroids or anti-convulsants.
13. Patient agrees to discontinue St. Johns Wort at least 5 days before starting dasatinib or erlotinib.
14. Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
15. The patient's O^2 saturation must be >92% on room air.
16. (Phase II only) - Patient has never received prior therapy with dasatinib, or erlotinib, or another epidermal growth factor receptor (EGFR) or Src family kinase (SFK) inhibitor.
17. (Phase I only) - Histological or unequivocal cytological proof of solid tumor malignancy.
18. (Phase I only) - At least one prior systemic chemotherapy or biological therapy for recurrent or metastatic solid tumor (i.e., this protocol therapy must be administered as second line or greater), ), except if there is no standard or experimental systemic therapy available. If no effective systemic agent is available for first line therapy, then patients may be enrolled on the phase I as first line therapy.
19. (Phase I only) - Prior radiotherapy is permitted (see exclusion criterion 4 for details on unallowable radiotherapy).
20. (Phase II only) - Histological or unequivocal cytological proof of NSCLC.
21. (Phase II only) - NSCLC that is appropriate for systemic therapy without curative intent: Stage IV, Stage IIIB with pleural effusion, or incurable recurrent disease after surgery or radiotherapy.
22. (Phase II only) - Zero to one line of prior systemic therapy for recurrent or metastatic NSCLC. Prior adjuvant chemotherapy or adjuvant biologic therapy for NSCLC is not included as a line of prior therapy if it was completed greater than 3 months prior to recurrence, provided that the patient has never received any EGFR or SFK inhibitors.
23. (Phase II only) - Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
24. (Phase II only) - Availability of tumor tissue that is at least adequate for EGFR mutational analysis. This can come from pre-existing paraffin blocks (from diagnostic biopsy or surgical resection) or patient may undergo a biopsy for research purposes.
25. (Phase II only) - Prior radiotherapy is permitted as long as there is measurable disease outside of the radiotherapy port OR clearly recurrent and growing within the radiotherapy port (see exclusion criterion 2 for details on unallowable radiotherapy).

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or have child-bearing potential and are unwilling/unable to use an acceptable method of contraception for the entire study period and for at least 4 weeks after cessation of the study drugs. All women of child-bearing potential must have a negative pregnancy test prior to first receiving protocol therapy. If the pregnancy test is positive, the patient must not receive dasatinib or erlotinib, and must not be enrolled on the study
2. Radiotherapy to ribs, sternum, pelvis, vertebrae or skull within 4 weeks prior to entering the study. (If none of these axial skeletal areas are included in the radiotherapy field, patients may have received palliative radiotherapy to long bones provided that it has ended at least 2 weeks prior to initiation of dasatinib-erlotinib therapy.)
3. Patients with any of the following cardiac problems should be excluded: (a) Uncontrolled angina, congestive heart failure, or myocardial infarction within the previous 6 months; (b) Diagnosed congenital long QT syndrome; (c) Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes); (d) Prolonged [1] corrected QT interval (QTc) interval on pre-entry electrocardiogram (> 450 msec in women or >440 msec in men). If the automated reading is prolonged, the ECG should be manually over read.
4. Continued from Exclusion #4: (e) Any history of second or third degree heart block unless they currently have a pacemaker; (f) Heart rate < 50 / minute on pre-entry electrocardiogram;(g) Uncontrolled hypertension defined as systolic blood pressure > 150 or diastolic >100;(h) Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration.
5. Patients with pericardial effusion > grade 1 (by Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0).
6. Patients with pleural effusion > grade 2 (by CTCAE v3.0). A grade 3 pleural effusion that is managed by a thoracentesis or an indwelling catheter is allowable as long as supplemental oxygen is not required.
7. Patients with any condition that impairs their ability to swallow, retain, or absorb dasatinib or erlotinib tablets are excluded. This includes any condition resulting in an inability to take oral medication, a requirement for IV alimentation, prior surgical procedures that have resulted in chronic malabsorption, or active peptic ulcer disease.
8. Patients with > grade 2 neuropathy
9. Patients with a history of pulmonary fibrosis (other than in a radiated field).
10. Patients with inflammatory bowel disease or uncontrolled chronic diarrhea.
11. Patients with a history of significant bleeding disorder unrelated to cancer, including: (a) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease); (b) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies); (c) Ongoing or recent (</= 3 months) significant gastrointestinal bleeding, defined as clinically evident hematemesis or hematochezia requiring therapeutic intervention.
12. Known HIV-positive patients are ineligible because of the potential for pharmacokinetic interactions between dasatinib and antiretroviral therapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
13. Pts currently receiving any of the following medications will be excluded: (a) Any concurrent systemic anticancer therapy; (b) Any concurrent investigational agents (c) Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Pts must discontinue such drugs 7 days or more prior to starting dasatinib):i. quinidine, procainamide, disopyramide;ii. amiodarone, sotalol, ibutilide, dofetilide;iii. erythromycin, clarithromycin;iv. chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
14. Continued from Exclusion#14:v.cisapride,bepridil,droperidol,methadone,arsenic, chloroquine,domperidone,halofantrine,levomethadyl,pentamidine,sparfloxacin, lidoflazine;(d)The concomitant use of H2 blockers or proton pump inhibitors w/ dasatinib is not recommended.The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in pts receiving dasatinib therapy.If antacid therapy is needed,the antacid dose should be administered at least 2 hours prior to or 2 hours after the dose of dasatinib.
15. Continued from Exclusion #15: (e)Pt may not be receiving any prohibited CYP3A4 inhibitors Potent inhibitors of CYP3A4 are prohibited during study; for such medications, a wash-out period of 7 days is required prior to starting dasatinib. Potent CYP3A4 inhibitors include: · itraconazole, ketoconazole, miconazole, voriconazole; amprenavir, atazanavir, fosamprenavir, indinavir, nelfinavir, ritonavir; ciprofloxacin, clarithromycin, diclofenac, doxycycline, enoxacin, imatinib, isoniazid, ketamine nefazodone, nicardipine, propofol, quinidine, telithromycin. (f) St.Johns Wort
16. The patient has received prior investigational therapy, chemotherapy, radiotherapy, or major surgery within 3 weeks of initiating study drug.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faye M. Johnson, MD, PhD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gold KA, Lee JJ, Harun N, Tang X, Price J, Kawedia JD, Tran HT, Erasmus JJ, Blumenschein GR, William WN, Wistuba II, Johnson FM. A phase I/II study combining erlotinib and dasatinib for non-small cell lung cancer. Oncologist. 2014 Oct;19(10):1040-1. doi: 10.1634/theoncologist.2014-0228. Epub 2014 Aug 28. PMID 25170013
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 6, 2008 to July 18, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 53 participants registered, only 47 were eligible and treated. The study was terminated early due to futility.
Groups:
- Dasatinib + Erlotinib: Dasatinib orally starting dose 70 mg/day & Erlotinib 150 mg orally/day every 21 day cycle.
Period: Overall Study
Arm/Group | Dasatinib + Erlotinib
Started | 47
Phase I | 12
Phase II | 35
Completed | 42
Not Completed | 5
Not completed — Disease Progression | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Dasatinib + Erlotinib: Phase I: Dasatinib orally starting dose 70 mg/day & Erlotinib 150 mg orally/day every 21 day cycle.
- Dasatinib + Erlotinib: Phase 2: MTD from Phase I Dasatinib orally dose 70 mg/day & Erlotinib 150 mg orally/day every 21 day cycle.
- Total: Total of all reporting groups
Arm/Group | Dasatinib + Erlotinib: Phase I | Dasatinib + Erlotinib: Phase 2 | Total
Number analyzed (Participants) | 12 | 35 | 47
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 74] | 63 [44 to 89] | 62 [44 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 17 | 21
  Male | 8 | 18 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 12 | 33 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 12 | 29 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 35 | 47

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerable Dose (MTD) of Dasatinib Given With Erlotinib Hydrochloride
Description: MTD defined as the highest dose level in which 6 patients have been treated with less than 2 instances of dose limiting toxicity (DLT). Dose-limiting toxicity (DLT) defined using NCI Common Terminology Common Terminology Criteria for Adverse Events (CTCAE) version 3 as: grade 3 or higher non-hematologic toxicity (excluding initial nausea and vomiting), grade 4 neutropenia, febrile neutropenia, or grade 4 thrombocytopenia. Grade 3-4 nausea and vomiting that cannot be controlled within 2 weeks with anti-emetics considered a DLT.
Time Frame: Baseline and at Day 21
Measure: Number; unit: mg/day
Arm/Group | Dasatinib + Erlotinib
Number analyzed (Participants) | 12
mg/day | 70

2. Secondary Outcome: Phase II: Number of Participant With Response According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. Patients who have a partial or complete response or stable disease are defined as progression free. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least 30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease (PD): At least 20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase.
Time Frame: 12 Weeks
Population: One participant only received one day of therapy therefore was not evaluable for efficacy analyses; a second participant discontinued study treatment.
Measure: Number; unit: participants
Groups:
- Dasatinib + Erlotinib: Dasatinib orally 70 mg/day & Erlotinib 150 mg orally/day every 21 day cycle.
Arm/Group | Dasatinib + Erlotinib
Number analyzed (Participants) | 33
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 5
  Progressive Disease (PD) | 13
  Stable Disease (SD) | 15

3. Secondary Outcome: Phase II: Progression-Free Survival (PFS) Rate
Description: A modified Thall, Simon, and Estey (1995) design used in the phase II study to monitor the proportion of patients with NSCLC who are alive and progression free (PFS) at twelve weeks after commencing treatment with dasatinib and erlotinib.
Time Frame: 12 Weeks
Population: Of the 35 participants in the Phase II portion of the study, one participant received one day of therapy therefore was not evaluable for efficacy analyses; a second participant discontinued study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dasatinib + Erlotinib
Number analyzed (Participants) | 33
Percentage of Participants | 53

ADVERSE EVENTS:
Time Frame: Adverse event collection was through each 3 week treatment cycle, up to 12 weeks of assessment with treatment.
Arm/Group | Dasatinib + Erlotinib
Serious Adverse Events (participants affected / at risk) | 3/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib + Erlotinib (N=47)
Death (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Multi-Organ Failure (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib + Erlotinib (N=47)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Acidosis (Metabolism and nutrition disorders) | 1 (2)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 3 (3)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 9 (10)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 11 (17)
Allergic rhinitis (Immune system disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 18 (20)
Anxiety (Nervous system disorders) | 7 (7)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 15 (23)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Auditory/Ear (Ear and labyrinth disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bilirubin increased (Metabolism and nutrition disorders) | 4 (8)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 24 (54)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (4)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac General (Cardiac disorders) | 2 (4)
Cardiac pain (Cardiac disorders) | 1 (1)
Cardiac troponin I increased (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 5 (6)
Chest wall pain (Cardiac disorders) | 1 (1)
Coagulation (Blood and lymphatic system disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis, infectious (Gastrointestinal disorders) | 1 (1)
Conjunctival disorder (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (20)
Constitutional Symptoms (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (34)
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 1 (1)
Creatinine increased (Metabolism and nutrition disorders) | 13 (26)
Dehydration (Gastrointestinal disorders) | 4 (4)
Depression (Psychiatric disorders) | 11 (11)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 32 (40)
Dizziness (Nervous system disorders) | 5 (5)
Dry eye syndrome (Eye disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 (64)
Edema limbs (General disorders) | 9 (10)
Electrocardiogram QTc interval prolonged (Cardiac disorders) | 1 (1)
Endocrine (Endocrine disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Fatigue (General disorders) | 38 (55)
Fever (Investigations) | 6 (7)
Flushing (Endocrine disorders) | 1 (1)
Gait abnormal (Musculoskeletal and connective tissue disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (4)
Gastrointestinal (Gastrointestinal disorders) | 4 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 12 (13)
Hearing loss (Ear and labyrinth disorders) | 3 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 34 (80)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 1 (1)
Hot flashes (Reproductive system and breast disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Cardiac disorders) | 9 (9)
Hypoparathyroidism (Endocrine disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Infection (Infections and infestations) | 3 (3)
Infection (Other) (Infections and infestations) | 3 (3)
INR increased (Blood and lymphatic system disorders) | 1 (1) — INR - International Normalized Ratio of prothrombin time
Insomnia (General disorders) | 8 (8)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (9)
Localized edema (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphatics (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 9 (34)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 11 (25)
Mini mental status examination abnormal (Psychiatric disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 5 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 30 (34)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neurology (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1)
Oral pain (General disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 14 (27)
Pain (Other) (General disorders) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes